CLINICAL TRIAL: NCT04414176
Title: Determining the Prevalence of Premature Coronary Heart Disease and it's Risk Factors According to Different Ethnicities and Religions in Iran and Developing a Biobank for Genetic and Epigenetic Studies
Brief Title: Iran- Premature Coronary Artery Disease
Acronym: I-PAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Iran Ministry of Health, Treatment, and Medical Education (Unknown)
Responsible Party: Principal Investigator, Ehsan Zarepur, Dr. Ehsan Zarepur (Cardiology resident, PhD candidate), Isfahan University of Medical Sciences
Other Study IDs: 296055
Record Dates: First submitted 2020-01-11; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Coronary Vessels
Keywords: Premature coronary heart disease; Ethnicity; Religion; Biobank

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be evaluated for fasting blood sugar and lipid profiles. All biological samples (serum, plasma, buffy coat, whole blood, urine, stool, and saliva) will be transferred to the central lab of the Isfahan Cardiovascular Research Institute to create a biobank (-80 c) for future genetic and epigenetic studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with coronary artery stenosis more than 75% (or left-main stenosis more than 50%) are defined as case group
- Control: Patients with normal angiography are considered as control group.

SUMMARY:
This case-control study will be conducted all over the country (in Persian, Kurd, Azari, Arab, Lor, Bakhtiari, Baluch, Turkman, Qashqai, Gilak and in Muslims, Christians, Jewish, and Zoroastrian). the investigators intend to recruit patients (men 60≥ years of age and women 70≥ years of age) who underwent coronary angiography. Patients with coronary artery stenosis more than 75% (or left-main stenosis more than 50%) are defined as case group and patients with normal angiography are considered as the control group. at the same time, the prevalence of premature coronary artery disease in patients with positive angiography will be calculated.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is one of the most important causes of mortality in the world and accounts for up to 30% of deaths. CHD is also prevalent in Iran and in some studies, the prevalence of the disease has been reported to be about 20 to 30 percent. The prevalence of premature coronary heart disease (CHD) is increasing every year, which is related to the risk factors for cardiovascular disease in humans. The prevalence of premature CHD in Iran is also high, which justify better understanding of the factors affecting it.

Many known risk factors are involved in coronary artery disease, including age, sex, obesity, high blood pressure, diabetes, dyslipidemia, smoking and family history. These risk factors do not have the same prevalence or attributable risk among different ethnicities and religions. Also due to genetic differences, the effect of environmental factors can accelerate or diminish the effects of some factors on the occurance of premature CHD. These mechanisms are often unknown, but high-risk environments can trigger an earlier onset of CHD in people who are genetically susceptible. This relation is called the genetic-environment interaction. As showed in previous reports, CHD is a multifactorial disease that can be affected by environmental factors and expression of different genes.

In this case-control study the investigators intend to recruit documented CHD patients who underwent coronary angiography from diverse ethnic and religious groups. A total of 5000 individuals from different ethnic backgrounds such as Persian (fars), Turk, Kurd, Arab, Lor, Bakhtiari, Baluch, Turkman, Qashqai, Gilak and in Muslims, Christians, Jews, and Zoroastrians will be selected throughout the country. Sampling among different ethnicities and religions will be based on their proportion of the total population.

Variables such as age, sex, ethnicity, religion, socioeconomic characteristics (educational level, working status, income), history of smoking, alcohol consumption, addiction, family and personal history of CHD, psychosocial habit, physical activity, and dietary habits will be collected. The heart rate and systolic and diastolic blood pressure will be taken twice in sitting position, and under standard conditions and the average of the two measurements will be recorded. The patient's weight (in kilograms), and height (in meters), the circumference of the wrist, neck, thigh, waist, and hip (all in centimeters) will be measured in light clothes and without shoes and body mass index and waist to hip ratio will be calculated.

Blood samples will be evaluated for fasting blood sugar and lipid profiles (Triglyceride, High-density lipoprotein-C, Low-density lipoprotein-C, and Total Cholesterol).

Samples of serum, plasma, buffy coat, whole blood, urine, stool, and saliva will be frozen and Individuals genetic and epigenetic variations will be examined in later stages.

All biological Samples will be transferred to the central lab of the Isfahan Cardiovascular Research Institute to create a BioBank for future genetic and epigenetic studies. The data collection teams will receive the necessary training in several sessions and the supervisory committee will regularly monitor the implementation of the plan.

ELIGIBILITY:
Inclusion Criteria:

* Men and women less than 60 and 70 years respectively
* Ethnicity
* Coronary artery stenosis more than 75% (or left-main stenosis more than 50%) or patients with normal angiography

Exclusion Criteria:

* patients with past medical history of CABG or documented coronary stenosis

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with documented coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-08-25 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Odds ratio | 2018 to 2020
  Odds ratio for life style risk factors among different ethnicities and religions

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan Cardiovascular Research Institute, Isfahan, Iran